CLINICAL TRIAL: NCT02722785
Title: PeRioperative Study of Exercise Training - a None-randomized Feasibility Study: Usual Care Observation vs Exercise Training Intervention in Patients With Operable Cancer of the Gastroesophageal Junction
Brief Title: PeRioperative Study of Exercise Training in Patients With Operable Cancer of the Gastroesophageal Junction
Acronym: PRESET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jesper Frank Christensen, PhD (Other)
Responsible Party: Sponsor-Investigator, Jesper Frank Christensen, PhD, PhD, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRESET - GEJ Cancer
Record Dates: First submitted 2016-03-10; First posted 2016-03-30 (Estimated); Last update posted 2018-08-15 (Actual); Status verified 2018-08

CONDITIONS: Gastro-esophageal Cancer
Keywords: Exercise training; Surgical complications; Cancer prognosis; Muscle function; Body composition; Pulmonary function; Quality of life

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual Care Observation Group (No Intervention): Patients allocated to usual care control will receive the standard patient care program as provided by the department of surgical gastroenterology, Rigshospitalet
- Aerobic and Resistance Exercise Training (Experimental): Patients allocated to this group will receive usual care plus a supervised aerobic and resistance exercise program at CFAS' facilities consisting of 2 weekly sessions of approximately 60 minutes.
  Interventions: Behavioral: Aerobic and Resistance Exercise Training

INTERVENTIONS:
Behavioral: Aerobic and Resistance Exercise Training — Supervised aerobic and resistance exercise program consisting of 2 weekly sessions of approximately 60 minutes. Patients will perform a test of maximum cardio-respiratory (Watt-max test) and muscle strength (1 repetition maximum [1-RM] test) capacity. Using the patient's individual capacity score (Watt-max and 1RM), a personalized exercise program will be prescribed. After a light warm-up, patients will perform 20-30 min of aerobic interval training of stationary bicycle. Resistance training comprises 4 exercises for the major muscle groups: chest press, leg press, lateral pull, and knee extension with 3-4 sets of 8 to 15 repetitions. Each session will be supervised by trained instructors to ensure proper technique, and progression in training load.
  Arms: Aerobic and Resistance Exercise Training

SUMMARY:
Background:

For patients diagnosed with operable cancer of the gastro-esophageal junction (GEJ), the perioperative course of therapy is associated with severe deconditioning which includes weight loss and poor physical function, which are strong predictor of post-surgical complication and survival . A strong rationale exists to explore how to develop supportive interventions aimed at maintaining/improving muscle function (lean body mass and muscle strength) during the pre-surgical phase.

This study explores the safety, feasibility and efficacy of structured pre- and post-operative exercise training in patient undergoing surgery for cancer of the gastro-esophageal junction.

Subjects: Patients with histologically verified, resectable adenocarcinoma of the GEJ scheduled for treatment af Rigshospitalet, Copenhagen, Denmark.

Methods: In a case-control design, patients will be allocated to either an exercise training intervention group, or a usual-care observational group, based on geographical location. Forty patients will be included in this case-control study and allocated by geographical region as follows; 20 training intervention-cases living in the greater Copenhagen area, and 20 observational control subjects living outside the greater Copenhagen area.

All patients will undergo a total of 5 assessments during the perioperative trajectory; twice prior to surgery (baseline and pre-surgery test), three post-surgery (2 week post- and 15 weeks post-surgery, and at 1-year follow-up).

Assessments include measures of body composition by DXA scan and bioelectrical impedance analysis: systemic inflammation in fasting blood sample; quality of life by self-report questionnaires; physical function by handgrip strength and sit-to-stand test.

As optional procedures, we will collect biological tissue from tumor, muscle and fat biopsies and a 10 ml blood sample at baseline and pre-surgery test only. Also, we will collect blood samples before, during and after an acute exercise bout exercise in order to explore the acute systemic changes in exercise-regulated biomarkers.

DETAILED DESCRIPTION:
BACKGROUND AND RATIONALE Patients diagnosed with operable cancer in upper gastro-intestinal (GI) tract undergo serious therapeutic procedures including invasive surgery combined with chemo- or chemo-radio therapy before (neo-adjuvant) and/or after (adjuvant) surgery. Despite recent advances, especially in surgical techniques and patient care follow-up, the population is faced with one of the worst prognosis for patients with operable staged disease, with a 5-year relative survival of 35-40%. The only possibility of long-term survival is positive surgical outcome, which includes the surgical principle of performing wide clearance, achieving a negative margin (R0 resection), and performing a radical lymphadenectomy. To this end, considerable efforts have been made in recent years optimizing the perioperative period in order to provide the patients and the surgeons with the best possible chances of achieving this surgical outcome.

Adenocarcinoma of the gastro-esophageal junction (GEJ) has increased in incidence over the last quarter century. For patients presenting with localized disease, advances in standards of care have emerged in recent years which have improved disease management. Firstly, comprehensive staging with Computed Tomography (CT), endoscopic ultrasound, diagnostic laparoscopy and fluoro deoxy glucose position emission tomography (18FDG-PET) permits exclusion of patients for curative therapy who might previously have been scheduled for resection. Secondly, evidence supports that esophagectomy is performed in high-volume hospitals by high-volume surgeons. Finally, standard neoadjuvant and adjuvant therapies are performed in most centers for patients with localized esophageal adenocarcinoma which has improved both short- and long-term cancer outcomes.

Prognostic role of Muscle Function in upper GI cancer For all upper GI cancers, including GEJ, the perioperative course of therapy is associated with severe deconditioning which includes weight loss and poor physical function. Over the last decade, strong observational evidence has emerged supporting that poor pre-surgical muscle function, defined as either low muscle mass/area (sarcopenia) or low functional strength, is a strong independent predictor of post-surgical outcomes including mortality, surgical complications and chemotherapy dose-reduction. Importantly, strong evidence across different malignancies has shown that the prognostic value of muscle function is independent from body mass, and may actually be under-reported due to sarcopenic obesity. Thus, current available therapeutic countermeasures in clinical practice, which exclusively involve nutritional interventions, may have limited potential for ameliorating the progressive muscle dysfunction during perioperative treatment for GEJ cancer.

Exercise-Oncology and Upper GI cancer Epidemiological evidence across both heterogeneous and homogeneous groups of cancer patients have shown that low physical activity level after diagnosis is associated with poor disease-specific and overall survival. Despite a general emerging interest, limited attention has been dedicated to the exploration of safety, feasibility and efficacy of structured exercise interventions in patients with upper GI cancer. However, data from recent studies suggests an unmet potential of physical exercise in these patients, with particular emphasis on the pre-surgical period.

STUDY OBJECTIVES Primary Objective

• To explore safety and feasibility of structured exercise in the pre- and post-operative phases among patients undergoing treatment for operable GEJ cancer

Secondary objectives:

* To explore the effect of perioperative exercise training on clinical (e.g. clindo-davien score, pneumonia, anastomotic leakage) physiological (e.g. muscle strength, physical function) and psycho-social (e.g. fatigue, emotional well-being, anxiety) endpoints relative to usual care.
* To explore the prognostic role of pathophysiological profile (physical function, pulmonary function, and body-composition) on post-surgical complications

Explorative objectives:

* To explore molecular adaptations of metabolism and physiology in tumor, muscle and fat samples taken before and after neo-adjuvant chemotherapy in the pre-operative phase in (a sub-group of) patients allocated to exercise training or usual care
* To explore the acute response in immune cells, hormones and cytokines in blood samples taken before, during and after a single exercise session
* Collection of blood and tissue samples for storage in bio-bank for future research.

STUDY DESIGN This prospective, regional-based case-controlled feasibility trial will include in a minimum of 40 patients, including 20 training intervention-cases who are residents in greater Copenhagen Area, and 20 usual care controls living outside the greater Copenhagen area.

Recruitment: Patients will be recruited from the department of surgical gastroenterology, Rigshospitalet, following multidisciplinary medical conference. The responsible physicians will provide oral information and present patients with the written information of the study.

Patients who are willing to participate will sign informed consent, before any study related procedures are performed. After signing informed consent, patients are scheduled for baseline assessment and will be allocated based on geographical location (home-town municipality), to one of two experimental arms:

I) Patient residing OUTSIDE the Copenhagen area, will be allocated to a usual care observation group, which includes nurse-based follow up procedures and information on life style factors (diet, smoking cessation, alcohol, and physical activity).

II) Patients residing WITHIN the Copenhagen area, will be allocated to usual care plus hospital-based aerobic and resistance training at Centre for Physical Activity Research, Rigshospitalet

Procedures will involve assessment-measures conducted a total of 5 times during the study period: twice prior to surgery (baseline and pre-surgery test), twice post-surgery (3 week post- and 15 weeks post-surgery) and at 1-year follow-up.

The following assessments will be performed:

1. Body composition by Bioelectrical Impedance
2. Fasting blood sample for analyses of plasma biochemistry (cholesterol, triglycerides, inflammatory markers, HbA1C)
3. Health related Quality of Life questionnaires
4. Physical function: Handgrip strength and sit-to-stand test.
5. Forced Expiration Volume in 1 second (FEV1)
6. Biological tissue sampling (OPTIONAL): tumor, muscle and fat biopsies and blood samples - only baseline and pre-surgery.
7. Acute Exercise Response (OPTIONAL); blood samples taken before and after a single exercise session.

ANALYTIC PLAN As a feasibility study, this trial is explorative in nature and performed primarily in order to determine whether it is appropriate to advance with a larger scaled randomized controlled trial.

Primary aim

Safety and feasibility of perioperative exercise training in patients with operable GEJ cancer

In order to evaluate the safety and feasibility of the pre- and post-surgical exercise in patients with operable cancer of the gastro-esophageal junction, incidence of serious adverse events in both groups will be determined, and adherence to exercise, assessed by number of training sessions completed in the training group.

Secondary aims

Efficacy of perioperative exercise training to improve clinical, physiological and psycho-social outcomes in patients operable GEJ cancer.

In order to determine whether exercise training has the capacity to improve study outcomes intragroup changes, and inter-group differences for study outcomes will be calculated. For this purpose a random effect analysis will be performed with repeated measures and study outcomes as dependent variables, with the covariates "group", "time" and their interaction as fixed effects, and a random effect of "patient", adjusted for baseline-score, chemotherapy regimen, and surgical procedure (conventional vs laparoscopic).

Prognostic role of pathophysiological profile in patients with operable GEJ cancer

In order to explore the prognostic role of the study assessment outcomes on key clinical endpoints: post-surgical complications, hospital stay duration and disease free and overall mortality risk over the first years after surgery, by a general linear regression models with clinical endpoints being the dependent variable, and study assessment outcomes as the independent variables adjusted for baseline-score, chemotherapy regimen, and surgical procedure (conventional vs laparoscopic). For each variable (physical function, pulmonary function, and body-composition), the predictive value of: I) the diagnostic level (prior to neo-adjuvant therapy), II) the pre-surgical level (after neo-adjuvant treatment) and III) the change score from diagnostic to pre-surgical level (during neo-adjuvant therapy) will be determined.

Dropouts and Missing Observations Patients who wish to drop-out of the study during the intervention-periods will be offered to remain in the study with regard to test-assessments. Patients who drop out prior to 'visit 2' will be replaced. For between-group analyses, all drop-outs and missing observations will be handled by the "missing at random" principle.

ETHICAL CONSIDERATIONS This study will be conducted in accordance with the regional ethical committee and the Declaration of Helsinki (1964) with its subsequent revisions. The protocol and any substantial amendments, the study patient information and consent form, as well as other relevant or requested material have been approved by the local ethics committee (Videnskabsetisk Komite) for the Capital Region of Denmark (Protocol number: H-15014904) and is reported to the Danish Data Protection Agency (Datatilsynet: RH-2016-33, I-Suite nr.: 04396) through Rigshospitalet/Capital Region of Denmark (j.nr. 2012-58-0004).

The project is expected to cause limited risks, side effects and discomfort. All procedures will be performed by experienced physicians, therapists and physiologists with relevant safety, and patients will not experience any kind of delays or complications related to treatment or control process due to participation in the project. Patients may at any time, and without justification, retract their consent.

ELIGIBILITY:
Inclusion Criteria:

Patients diagnosed with histologically verified, resectable adenocarcinoma of the GEJ.

Exclusion Criteria:

* Deemed in-operable at multidisciplinary medical conference
* Pregnancy
* Any other known malignancy requiring active treatment
* In-eligible to chemotherapy
* Performance status > 1
* Physical disabilities precluding physical testing and/or exercise
* Inability to read and understand Danish

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-04 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Incidence of Adverse Events (AEs) and Serious Adverse Events (SAEs) | Baseline to 1-year follow-up
  Recording of adverse events will be separated into two procedures: recordings during trial visits and recordings during exercise sessions.
  AE/SAE recording during trial assessment visits This procedure will concern any AE/SAE which can be attributed to study-related assessment procedures during the trial visits, i.e. discomfort during physical tests or blood sampling, which will be recorded immediately during the visit and recorded for the given visit. Also, for each trial visit we will collect patients' self-report of AE/SAEs, which may have occurred during the period since the last trial visit without our knowledge.
  AE/SAE recording during exercise sessions For every exercise session, a trained instructor will supervise the exercise program including recording of AE/SAEs during these session
Adherence to prescribed exercise program | Baseline to 3 months post surgery
  Proportion of exercise sessions completed.

SECONDARY OUTCOMES:
Changes in fat percentage | Baseline to 1-year follow-up
  Body fat percentage is assessed measuring bioelectrical impedance in the body using a state-of-the-art Bioelectrical Impedance Analyzer (Tanita MC-780 MA, Tokyo, Japan). The degree of difficulty with which electricity passes through a substance is known as the electrical resistance, and the percentage of fat and other body constituents can be inferred from measurements of this resistance. The analyzer measures body composition using a constant current source with a high frequency current (50kHz, 90µA) with 8 electrodes positioned so that electric current is supplied from the electrodes on the tips of the toes of both feet, and voltage is measured on the heel of both feet. The current flows into the upper limbs or lower limbs, depending on the body part(s) to be measured. Patients with pacemakers or other electrical implants will not undergo this measure due to safety specifications.
Changes in lean mass | Baseline to 1-year follow-up
  Lean mass is assessed measuring bioelectrical impedance in the body using a state-of-the-art Bioelectrical Impedance Analyzer (Tanita MC-780 MA, Tokyo, Japan). The degree of difficulty with which electricity passes through a substance is known as the electrical resistance, and the percentage of fat and other body constituents can be inferred from measurements of this resistance. The analyzer measures body composition using a constant current source with a high frequency current (50kHz, 90µA) with 8 electrodes positioned so that electric current is supplied from the electrodes on the tips of the toes of both feet, and voltage is measured on the heel of both feet. The current flows into the upper limbs or lower limbs, depending on the body part(s) to be measured. Patients with pacemakers or other electrical implants will not undergo this measure due to safety specifications.
Changes in fat mass | Baseline to 1-year follow-up
  Body fat mass is assessed measuring bioelectrical impedance in the body using a state-of-the-art Bioelectrical Impedance Analyzer (Tanita MC-780 MA, Tokyo, Japan). The degree of difficulty with which electricity passes through a substance is known as the electrical resistance, and the percentage of fat and other body constituents can be inferred from measurements of this resistance. The analyzer measures body composition using a constant current source with a high frequency current (50kHz, 90µA) with 8 electrodes positioned so that electric current is supplied from the electrodes on the tips of the toes of both feet, and voltage is measured on the heel of both feet. The current flows into the upper limbs or lower limbs, depending on the body part(s) to be measured. Patients with pacemakers or other electrical implants will not undergo this measure due to safety specifications.
Changes in Plasma Total-Cholesterol concentrations | Baseline to 1-year follow-up
  Concentrations of total cholesterol will be measured in fasting blood samples by standard laboratory methods.
Changes in Plasma LDL-Cholesterol concentrations | Baseline to 1-year follow-up
  Concentrations of LDL-cholesterol will be measured in fasting blood samples by standard laboratory methods.
Changes in Plasma HDL-Cholesterol concentrations | Baseline to 1-year follow-up
  Concentrations of HDL-cholesterol will be measured in fasting blood samples by standard laboratory methods.
Changes in Plasma triglyceride concentrations | Baseline to 1-year follow-up
  Concentrations of triglyceride will be measured in fasting blood samples by standard laboratory methods.
Changes in HbA1C (fasting blood samples) | Baseline to 1-year follow-up
  HbA1C will be measured in fasting blood samples by standard laboratory methods.
Changes in Tumor Nekrosis Factor alpha (TNFa) concentration | Baseline to 1-year follow-up
  Concentrations of TNFa will be measured in fasting blood samples by Enzyme-linked immunosorbent assay (ELISA) analyses.
Changes in Interleuken (IL)-6 concentration | Baseline to 1-year follow-up
  Concentrations of IL-6 will be measured in fasting blood samples by Enzyme-linked immunosorbent assay (ELISA) analyses.
Changes in Interleukin (IL)-8 concentration | Baseline to 1-year follow-up
  Concentrations of IL-8 will be measured in fasting blood samples by Enzyme-linked immunosorbent assay (ELISA) analyses.
Changes in Interleukin (IL)-10 concentration | Baseline to 1-year follow-up
  Concentrations of IL-10 will be measured in fasting blood samples by Enzyme-linked immunosorbent assay (ELISA) analyses.
Changes in patient-reported Quality of Life - FACT | Baseline to 1-year follow-up
  Patient reported quality of life is measured by Functional Assessment of Cancer Treatment (FACT)
Changes in Sleep Quality | Baseline to 1-year follow-up
  Patient reported sleep quality is measured by the Pittsburgh Sleep Quality Index (PSQI) questionaire
Changes in Anxiety and Depression | Baseline to 1-year follow-up
  Patient reported Anxiety and Depression is measured by the Hospital Anxiety and Depression Scale (HADS).
Changes in Physical Activity level | Baseline to 1-year follow-up
  Patient reported physical activity is measured by the Internations Physical Activity Questionaire (IPAQ) - short form
Changes in physical function | Baseline to 1-year follow-up
  Sit-to-stand test: Lower-body physical function is assessed by 30-second sit-to-stand test. Using a chair fixed to the ground with a seat 45 cm above the ground subjects will be instructed to sit in the middle of the chair, back straight, arms crossed over their chest, feet flat on the floor. Correct technique will be demonstrated first, and subjects will practice for two-three repetitions. On the signal "go" subjects will be asked to stand then return to the seated position, as many times as possible in 30 seconds.
Changes in hand-grip strength | Baseline to 1-year follow-up
  Handgrip strength is assessed by hand-held dynamometer. Grip strength is measured in a seated position with the elbow flexed at 90°, with three attempts performed for each hand. During testing, the participant will be encouraged to exhibit the best possible force, and the best measure in the strongest hand will be used as test score.
Changes in Forced Expiration Volume in 1 second (FEV1) | Baseline to 1-year follow-up
  FEV1 is evaluated by validated assessment measure of pulmonary function. The patient is instructed to make a complete inspiration and then inserts the mouthpiece into the mouth, closes the lips around it but with the jaws apart, and blows out through the mouth as hard and as completely as possible with strong verbal encouragement given throughout this sequence. The FEV1 score is the fraction of the total volume which is expired in the first second

OTHER OUTCOMES:
Tissue sampling - Optional | At baseline and at surgery
  For the pre-surgical period (at baseline- and during surgery), we will ask for patients' separate consent to do a gastroscopy with sampling of a tumor biopsy; a muscle biopsy from m. vastus lateralis, fat biopsy from subcutaneous abdominal adipose tissue; and a blood sample, all of which will be collected during full anesthesia. A gastroscopy will be performed and endoluminal tumor biopsies will be collected under full anesthesia in patients who have given informed consent, after the diagnostic laparoscopy is completed. Muscle biopsies of approx. 200 mg per biopsy, will be collected from m. vastus lateralis using the Bergstrom-technique, and fat biopsies of approx. 200 mg per biopsy will be collected from the subcutaneous adipose tissue in the abdomen. Standard procedure requires the resection specimen to be dissected and cut open to determine lymph node classification and resection margins.

CONTACTS AND LOCATIONS:
Overall Officials: Jesper F Christensen, PhD, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Simonsen C, Thorsen-Streit S, Sundberg A, Djurhuus SS, Mortensen CE, Qvortrup C, Pedersen BK, Svendsen LB, de Heer P, Christensen JF. Effects of high-intensity exercise training on physical fitness, quality of life and treatment outcomes after oesophagectomy for cancer of the gastro-oesophageal junction: PRESET pilot study. BJS Open. 2020 Oct;4(5):855-864. doi: 10.1002/bjs5.50337. Epub 2020 Aug 28. PMID 32856785